CLINICAL TRIAL: NCT06823102
Title: Brain Connectivity Analysis to Predict Post Stroke Outcomes Following Traditional and Enhanced Neurorehabilitation by Transcranial Direct Current Stimulation and Anti-inflammatory Biomimetic Nanoparticles
Brief Title: Brain Connectivity Analysis
Acronym: Neurehab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP 22/24
Record Dates: First submitted 2025-01-29; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Neural Injury
Keywords: Non Invasive Brain Stimulation; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tDCS+standard rehabilitation (Experimental)
  Interventions: Other: tDCS
- tDCS sham+standard rehabilitation (Sham Comparator)
  Interventions: Other: tDCS
- standard rehabilitation (No Intervention)

INTERVENTIONS:
Other: tDCS — Transcranial direct current stimulation
  Arms: tDCS sham+standard rehabilitation; tDCS+standard rehabilitation

SUMMARY:
Stroke remains the leading cause of permanent disability. The neuromodulation technique of transcranial Direct Current Stimulation (tDCS) has the potential to serve as an adjuvant therapy to enhance neuronal connectivity following stroke. By combining electroencephalography (EEG) and tDCS, this study aims to investigate changes in network connectivity and cerebral plasticity, which are key factors in functional recovery after stroke.

The objectives are to: 1) analyze how tDCS modulates neuronal activity, 2) evaluate persistent effects in follow-up assessments, and 3) predict patient outcomes. Studies on human subjects will be complemented by research in a mouse model of stroke to: 1) identify the molecular mechanisms underlying tDCS effects on functional recovery, 2) establish correlations among functional, molecular, and connectivity indices, and 3) assess the efficacy of biomimetic nanoparticles in targeting injured brain tissue to reduce inflammation, enhance neuronal plasticity, and support functional recovery.

ELIGIBILITY:
Inclusion Criteria:

Age 18-90

* First ischemic stroke occurring 3-30 days after onset
* Residual upper limb function
* Ability to provide informed consent and understand instructions

Exclusion Criteria:

* Severe spasticity (Ashworth >2)
* Presence of additional neurological diseases
* Significant comorbidities
* History of intracerebral hemorrhage
* Severe neglect
* Contraindications to tDCS

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Evaluate effects of tDCS in short-term follow-ups in terms of EEG Coherence | from month 8 to month 12
  Analysis of Magnitude Squared Coherence to evaluate short-term tDCS effects
Evaluate persistent effect of tDCS in long-term follow-ups of EEG Coherence | From month 15 to the end of project
  Analysis of Magnitude Squared Coherence evaluate long-term tDCS effects
Evaluate effects of tDCS in short-term follow-ups in terms of EEG Connectivity | from month 8 to month 12
  Analysis of EEG Connectivity to evaluate short-term tDCS effects
Evaluate persistent effect of tDCS in long-term follow-ups of EEG Connectivity | From month 15 to the end of project
  Analysis of EEG Connectivity to evaluate long-term tDCS effects
Predict patients' outcome | through study completion, an average of 1 year
  Use of AI to predict the outcome of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Casa di cura San Raffaele Pisana, Rome, Rome, Italy